CLINICAL TRIAL: NCT03222076
Title: An Open-Label Preoperative Pilot Study Evaluating Nivolumab (Anti-PD-1 Antibody) Alone Versus Nivolumab Plus Ipilimumab (Anti-CTLA-4 Antibody) in Patients With Resectable (HCC)
Brief Title: Nivolumab With or Without Ipilimumab in Treating Patients With Resectable Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0097; NCI-2018-01106 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0097 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma; Resectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 2 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo liver surgery on day 1 of week 7. Beginning 4 weeks after surgery, patients continue nivolumab IV over 30 minutes every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab
- Arm B (ipilimumab, nivolumab) (Experimental): Patients receive ipilimumab IV over 90 minutes on day 1 and nivolumab as Arm A. Treatment repeats every 2 weeks for up to 3 cycles for nivolumab in the absence of disease progression or unacceptable toxicity. Patients undergo liver surgery on day 1 of week 7. Beginning 4 weeks after surgery, patients receive ipilimumab IV over 90 minutes every 6 weeks and nivolumab IV over 30 minutes every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm B (ipilimumab, nivolumab)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies the side effects and how well nivolumab with or with ipilimumab works in treating patients with liver cancer that can be removed by surgery. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
Primary Objective:

--To evaluate the safety and tolerability of therapy with nivolumab alone or nivolumab + ipilimumab in resectable HCC in the context of presurgical therapy.

Note: Note: As of January 8, 2020, 30 patients have been enrolled and 27 patients have been randomized. The PI decided to stop enrollment since the study has reached its target enrollment of 30 patients

Secondary Objectives:

--To assess the efficacy of presurgical nivolumab alone or nivolumab + ipilimumab therapy in HCC by estimating the objective response rate (ORR) and time to progression (TTP) per RECIST 1.1 progression-free survival (PFS).

Exploratory Objectives:

--To assess the immunological/biomarker changes in tumor tissues and peripheral blood in response to nivolumab alone or nivolumab + ipilimumab in HCC therapy (pre- vs post-treatment), and explore any potential association between these biomarker measures and antitumor response and immune-related response criteria (iRC) assessed by MD Anderson Department of Diagnostic Imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must give written informed consent prior to initiation of therapy, in keeping with the policies of the institution. Patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with the therapy.

   Target population
2. Patients with histologically confirmed HCC (Documentation of original biopsy for diagnosis is acceptable if tumor tissue is unavailable) or clinical diagnosis by AASLD criteria in cirrhotic subjects is required (presence of arterial hypervascularity with venous washout). For subjects without cirrhosis, histological confirmation is mandatory. The determination of resectability status will ultimately lie in the clinical judgment of the surgical oncologist and medical oncologist involved in the care of the patient.
3. Patient must have measurable disease defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) and measures ≥ 15 mm with conventional techniques or ≥ 10 mm with more sensitive techniques such as MRI or spiral CT scan.
4. Patient can have had prior treatment for HCC including prior surgery, radiation therapy, local-regional therapy (abalation or arterial directed therapies), and systemic therapy including sorafenib or chemotherapy (but not anti-PD-1 or anti-CTLA-4 therapy)
5. ECOG performance status ≤ 1.
6. Within 14 days of the first dose of study drug, patients must have adequate organ and marrow function as defined below:

   * Absolute neutrophil count ≥ 1,500/μL
   * Platelets ≥100,000/μL
   * Hgb > 9.0 g/dL (may be transfused or receive epoetin alfa [e.g., Epogen®] to maintain or exceed this level)
   * Total bilirubin ≤ 1.5 mg/dl
   * Serum creatinine ≤ 1.5 times the upper limit of normal or estimated CrCL >40mL/min.
   * AST (SGOT) and/or ALT (SGPT) ≤ 5 X institutional upper limit of normal Age and Sex
7. Men and women ≥ 18 years of age
8. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
9. Women must not be breastfeeding
10. WOCBP must agree to follow instructions for method(s) of contraception from the time of enrollment for the duration of treatment with study drug (s) plus 5 half-lives of study drug (s) plus 30 days (duration of ovulatory cycle) for a total of 5 months post treatment completion.
11. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug (s) plus 5 half-lives of study drug (s) plus 90 days (duration of sperm turnover) for a total of 7 months post-treatment completion.
12. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, WOCBP must still undergo pregnancy testing as described in these sections.

Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% per year when used consistently and correctly.

At a minimum, subjects must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective as listed below:

HIGHLY EFFECTIVE METHODS OF CONTRACEPTION

* Male condoms with spermicide
* Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena by WOCBP subject or male subject's WOCBP partner.
* Nonhormonal IUDs, such as ParaGard
* Tubal ligation
* Vasectomy
* Complete Abstinence* *Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs. Abstinence is only acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (eg, calendar, ovulation, symptothermal, profession of abstinence for entry into a clinical trial, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Subjects who choose complete abstinence are not required to use a second method of contraception, but female subjects must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence.

LESS EFFECTIVE METHODS OF CONTRACEPTION

* Diaphragm with spermicide
* Cervical cap with spermicide
* Vaginal sponge
* Male Condom without spermicide*
* Progestin only pills by WOCBP subject or male subject's WOCBP partner
* Female Condom* *A male and female condom must not be used together

Exclusion Criteria:

Any of the following criteria will disqualify the patient from participation:

Target Disease Exceptions

1. Any other malignancy from which the patient has been disease-free for less than 2 years, except for non-melanoma skin cancer, or in situ carcinoma of any site.

   Medical History and Concurrent Disease
2. Patients who have organ allografts.
3. Patients who have had a major surgical procedure, open biopsy, or significant traumatic injury with poorly healed wound within 6 weeks prior to first dose of study drug; or anticipation of need for major surgical procedure during the course of the study (other than defined by protocol); fine needle aspirations or core biopsies within 7 days prior to first dose of study drug. NOTE: Patients will be allowed to start cycle 1 day 1 therapy after 24 hours from pre-treatment biopsy.
4. Autoimmune disease: Patients with a history of inflammatory bowel disease (including crohn's disease and ulcerative colitis) are excluded from this study as are patients with a history of autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., wegener's granulomatosis]).
5. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
6. Any underlying medical condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea.
7. Patients who have had a history of acute diverticulitis, abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, GI obstruction, abdominal carcinomatosis which are known risks factors for bowel perforation, should be excluded from the study.
8. Patients who have a primary brain tumor (excluding meningiomas and other benign lesions), any brain metastases, leptomeningeal disease, seizure disorders not controlled with standard medical therapy, or history of stroke within the past year.
9. History of serious systemic disease, including myocardial infarction or unstable angina within the last 12 months, history of hypertensive crisis or hypertensive encephalopathy, uncontrolled hypertension (blood pressure of >140/90 mmHg) at the time of enrollment, New York Heart Association (NYHA) Grade II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (patients with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible), significant vascular disease or symptomatic peripheral vascular disease.
10. Patients who have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
11. Patients who are on high dose steroid (e.g. > 10 mg prednisone daily or equivalent) or other more potent immune suppression medications (e.g. infliximab)
12. Patients who have had influenza, hepatitis, or other vaccines within a month prior to initiation of study drugs.
13. Patients who have clinical history of coagulopathy, bleeding diathesis or thrombosis within the past year.
14. Patients who have serious, non-healing wound, ulcer, or bone fracture.
15. Pregnancy (positive pregnancy test) or lactation.
16. Patients with prior orthotropic liver transplantation.
17. Patients with cirrhosis and severe synthetic liver dysfunction (Child Pugh B-C).

    Prohibited Therapies and/or Medications
18. Patients must not have received prior anticancer therapy with anti-CLTA-4 or anti-PD1 for HCC. Patients receiving any concomitant systemic therapy for HCC are excluded.
19. Patients must not be scheduled to receive another experimental drug while on this study.
20. Patients who require ongoing anticoagulation will be excluded. Only aspirin will be permitted. Pre and post-surgical prophylactic anti-coagulation treatment is permitted.
21. Patients must not require total parenteral nutrition with lipids.

    Other Exclusion Criteria:
22. Any patients who cannot be compliant with the appointments required in this protocol must not be enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed O Kaseb, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kaseb AO, Hasanov E, Cao HST, Xiao L, Vauthey JN, Lee SS, Yavuz BG, Mohamed YI, Qayyum A, Jindal S, Duan F, Basu S, Yadav SS, Nicholas C, Sun JJ, Singh Raghav KP, Rashid A, Carter K, Chun YS, Tzeng CD, Sakamuri D, Xu L, Sun R, Cristini V, Beretta L, Yao JC, Wolff RA, Allison JP, Sharma P. Perioperative nivolumab monotherapy versus nivolumab plus ipilimumab in resectable hepatocellular carcinoma: a randomised, open-label, phase 2 trial. Lancet Gastroenterol Hepatol. 2022 Mar;7(3):208-218. doi: 10.1016/S2468-1253(21)00427-1. Epub 2022 Jan 20. PMID 35065057
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 excluded: 1 did not meet inclusion criteria; 2 declined to participate
  The study was amended in June 2019 to remove/exclude the enrollment of Arm C .
Groups:
- Arm A: Nivolumab: Nivolumab at 240 mg IV every 2 weeks for 3 doses followed by liver imaging and hepatic resection on day 1 of week 7, followed (after 4 weeks from surgery) by nivolumab 480 mg IV every 4 weeks in the adjuvant setting until disease progression or for 2 years, whichever is sooner
  Nivolumab: Given IV
- Arm B: Nivolumab Plus Ipilimumab: Nivolumab 240 mg IV every 2 weeks for 3 doses plus ipilimumab 1 mg/kg IV on day 1 of therapy (3 doses of nivolumab, 1 dose of ipilimumab) followed by hepatic resection followed (after 4 weeks from surgery) by nivolumab 480 mg IV every 4 weeks plus ipilimumab 1 mg/kg IV every 6 weeks to 4 doses in the adjuvant settingIpilimumab: Given IV
  Nivolumab: Given IV Ipilimumab: Given IV
- Arm C: Nivolumab Plus Ipilimumab: Nivolumab 240 mg IV every 2 weeks for 3 doses plus ipilimumab 1 mg/kg IV on day 1 of therapy (3 doses of nivolumab, 1 dose of ipilimumab; 6 weeks) in Unresectable patients followed by post-treatment biopsy
Period: Overall Study
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Ipilimumab | Arm C: Nivolumab Plus Ipilimumab
Started | 13 | 14 | 0
Completed | 13 | 14 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 2 of the patients (1 in the Nivolumab arm and 1 in the Nivolumab + Ipilimumab arm) was not included in the analysis of PFS because their surgical cancellations were unrelated to progressive disease.
Groups:
- Arm A: Nivolumab: Nivolumab at 240 mg IV every 2 weeks for 3 doses followed by liver imaging and hepatic resection on day 1 of week 7, followed (after 4 weeks from surgery) by nivolumab 480 mg IV every 4 weeks in the adjuvant setting until disease progression or for 2 years, whichever is sooner
- Arm B: Nivolumab Plus Ipilimumab: Nivolumab 240 mg IV every 2 weeks for 3 doses plus ipilimumab 1 mg/kg IV on day 1 of therapy (3 doses of nivolumab, 1 dose of ipilimumab) followed by hepatic resection followed (after 4 weeks from surgery) by nivolumab 480 mg IV every 4 weeks plus ipilimumab 1 mg/kg IV every 6 weeks to 4 doses in the adjuvant setting
- Total: Total of all reporting groups
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Ipilimumab | Arm C: Nivolumab Plus Ipilimumab | Total
Number analyzed (Participants) | 13 | 14 | 0 | 27
Age, Continuous [Median (Full Range); unit: years] | 64 [56 to 68] | 62 [53 to 72] |  | 64 [53 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 |  | 8
  Male | 11 | 8 |  | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 4 | 3 |  | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 3 | 4 |  | 7
  White | 6 | 7 |  | 13
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 14 |  | 27

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Presurgical Nivolumab With or Without Ipilimumab, Defined as the Number of Participants With of Adverse Events.
Description: The frequency of adverse events, serious adverse events (grade ≥3), and laboratory abnormalities. Graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Safety will be recorded through the incidence of adverse events, serious adverse events and specific laboratory abnormalities (worst grade) in each treatment arm.
Time Frame: Up to 5 years
Population: Cohort C that was discontinued due to non-accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Ipilimumab | Arm C: Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 13 | 14 | 0
Participants | 13 | 14 | 0

2. Secondary Outcome: Objective Response Rate
Description: Overall response rate, defined as the proportion of patients with a complete response or partial response after 6 weeks of therapy by RECIST 1.1 criteria divided by the number of randomly assigned patients.
Time Frame: After 6 weeks of therapy, up to 5 years
Population: Cohort C that was discontinued due to non-accrual.
Measure: Number; unit: participants
Groups:
- Arm C (Ipilimumab, Nivolumab): Patients receive ipilimumab and nivolumab as in Arm B. Patients undergo post-treatment biopsy on day 1 of week 7, then receive ipilimumab IV over 90 minutes every 6 weeks and nivolumab IV over 30 minutes every 4 weeks for up to 3 additional cycles in the absence of disease progression or unacceptable toxicity. Beginning 4 weeks after surgery, patients receive ipilimumab IV over 90 minutes every 6 weeks and nivolumab IV over 30 minutes every 4 weeks up to 2 years in the absence of disease progression or unacceptable toxicity.
  Ipilimumab: Given IV
  Nivolumab: Given IV
Arm/Group | Arm A (Nivolumab) | Arm B (Ipilimumab, Nivolumab) | Arm C (Ipilimumab, Nivolumab)
Number analyzed (Participants) | 13 | 14 | 0
participants | 3 | 0 |

3. Secondary Outcome: Time to Progression
Description: Time to progression defined as the time from the start of the study drug to the first documented tumor progression or recurrence of the tumor as determined by the investigator by RECIST 1.1 or immune-related response criteria.
Time Frame: Up to 5 years
Population: 2 of the patients (1 in the Nivolumab arm and 1 in the Nivolumab + Ipilimumab arm) was not included in the analysis of PFS because their surgical cancellations were unrelated to progressive disease.
  Upper limit of 95% Confidence Interval is not estimable due to insufficient number of participants and number of events.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Nivolumab) | Arm B (Ipilimumab, Nivolumab) | Arm C (Ipilimumab, Nivolumab)
Number analyzed (Participants) | 12 | 13 | 0
months | 9.4 [1.47 to NA] — 2 of the patients (1 in the Nivolumab arm and 1 in the Nivolumab + Ipilimumab arm) was not included in the analysis of PFS because their surgical cancellations were unrelated to progressive disease. | 19.53 [2.33 to NA] — 2 of the patients (1 in the Nivolumab arm and 1 in the Nivolumab + Ipilimumab arm) was not included in the analysis of PFS because their surgical cancellations were unrelated to progressive disease. |

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival, defined as the time from the start of treatment to the date of progessive disease, recurrence, or death, whichever occurred first. The Kaplan-Meier method will be used to estimate probability of PFS for each treatment arm.
Time Frame: Up to 5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Nivolumab) | Arm B (Ipilimumab, Nivolumab) | Arm C (Ipilimumab, Nivolumab)
Number analyzed (Participants) | 12 | 13 | 0
months | 9.4 [1.47 to NA] — 2 of the patients (1 in the Nivolumab arm and 1 in the Nivolumab + Ipilimumab arm) was not included in the analysis of PFS because their surgical cancellations were unrelated to progressive disease. | 19.53 [2.33 to NA] — 2 of the patients (1 in the Nivolumab arm and 1 in the Nivolumab + Ipilimumab arm) was not included in the analysis of PFS because their surgical cancellations were unrelated to progressive disease. |

ADVERSE EVENTS:
Time Frame: Overall Study (Up to 5 years)
Groups:
- Nivolumab: Nivolumab at 240 mg IV every 2 weeks for 3 doses followed by liver imaging and hepatic resection on day 1 of week 7, followed (after 4 weeks from surgery) by nivolumab 480 mg IV every 4 weeks in the adjuvant setting until disease progression or for 2 years, whichever is sooner
  Nivolumab: Given IV
- Nivolumab Plus Ipilimumab: Nivolumab 240 mg IV every 2 weeks for 3 doses plus ipilimumab 1 mg/kg IV on day 1 of therapy (3 doses of nivolumab, 1 dose of ipilimumab) followed by hepatic resection followed (after 4 weeks from surgery) by nivolumab 480 mg IV every 4 weeks plus ipilimumab 1 mg/kg IV every 6 weeks to 4 doses in the adjuvant settingIpilimumab: Given IV
  Nivolumab: Given IV Ipilimumab: Given IV
Arm/Group | Nivolumab | Nivolumab Plus Ipilimumab
All-Cause Mortality (participants affected / at risk) | 0/13 | 4/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 10/13 | 12/14
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab (N=13) | Nivolumab Plus Ipilimumab (N=14)
Anaemia (Investigations) | 2 (2) | 3 (3)
Increased alanine aminotransferase (Investigations) | 3 (3) | 7 (7)
Increased aspartate aminotransferase (Investigations) | 3 (3) | 7 (7)
Decreased platelet count (Investigations) | 2 (2) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 6 (6)
Hypothyroidism (Endocrine disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT03222076/Prot_SAP_000.pdf